CLINICAL TRIAL: NCT05245240
Title: Novel Inhibitors of Lipolysis in the Treatment of Lipid a Glucose Metabolism in Obstructive Sleep Apnea Syndrome
Acronym: NORRIS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Jan Polak, Principal Investigator, Faculty Hospital Kralovske Vinohrady
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NU21-01-00259
Record Dates: First submitted 2022-02-03; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Obstructive Sleep Apnea; Obesity
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity | interventions — Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Severe OSA group (Experimental): Dietary and physical activity intervention
  Interventions: Procedure: Dietary and physical intervention
- Mild OSA group (Experimental): Dietary and physical activity intervention
  Interventions: Procedure: Dietary and physical intervention

INTERVENTIONS:
Procedure: Dietary and physical intervention — Low-caloric diet (energy deficit 600 kcal/day based on indirect calorimetry measurements), individually tailored by a nutritional specialist according to patients' individual food preferences.
  Mild to moderate intensity exercise of aerobic/endurance type, performed 3 times a week for 30-90 minutes.

SUMMARY:
Obstructive sleep apnea syndrome (OSA) represents highly prevalent (typically overlooked, undiagnosed and untreated) disorder significantly increasing cardiovascular, cancer and overall mortality as well as increasing the risk of Type 2 diabetes and liver steatohepatitis. Unfortunately, adherence to state-of-the-art therapy with continuous positive airway pressure devices (CPAP) is poorly tolerated by patients, rendering a significant proportion (~60-70 %) of them at undiminished cardiovascular and metabolic risk warranting development of innovative, pharmacological, treatment options.

The overarching theme of this project is that metabolic impairments associated with OSA (e.g. Type 2 diabetes mellitus and non-alcoholic steatohepatitis) are causally mediated by elevated levels of circulating free fatty acids (FFA) originating from hypoxia-induced adipose tissue lipolysis. Increased plasma FFA subsequently induce insulin resistance, β-cell dysfunction, increase hepatic glucose output and stimulate lipid storage in liver. The investigators recently proved that hypoxia represents a powerful stimulus for adipocyte lipolysis and that experimental pharmacological inhibition of lipolysis prevented development of Type 2 diabetes in a mouse model of OSA. The goal of the project is to understand adipose tissue lipolysis derangements in OSA subjects and to evaluate the feasibility of lifestyle intervention as a mean to reduce spontaneous lipolysis.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a common condition affecting 5-15% of the general population characterized by a repetitive collapse of the upper airway during sleep. The ensuing apneas and hypopneas lead to episodic drops in oxyhemoglobin saturation (intermittent hypoxia) and recurrent arousals from sleep. Research over the last decade has demonstrated that OSA is independently associated with insulin resistance, glucose intolerance, type 2 diabetes mellitus (T2DM) and non-alcoholic steatohepatitis (NASH), however, molecular mechanisms mediating this causal link remain unknown. Increased sympathetic autonomic activity, alterations in corticotropic function, augmented oxidative stress and activation of inflammatory pathways represent possible intermediate mechanisms.

Research interest of the investigators is to explore the role of enhanced adipose tissue lipolysis and circulating free fatty acid (FFA) levels as a causal factor impairing metabolic homeostasis in OSA. The investigators as well as other researchers demonstrated that exposure to sustained and intermittent hypoxia increased adipocyte lipolysis in-vitro and in mice.

Enhanced spontaneous lipolysis in subcutaneous adipose tissue with subsequent FFA release into circulation is a predominant source of plasma FFA in obese and insulin resistant subjects. Plasma FFA levels subsequently provide energy for working muscle, however, it has been also recognized that FFA mediate important regulatory and endocrine functions. Indeed, obese individuals as well as T2DM patients are often characterized by higher FFA in plasma and elevated FFA levels are considered to be a causal factor inducing insulin resistance in muscle and liver and hampering insulin secretion and β-cells ultimately contributing to the development of Type 2. diabetes mellitus (T2DM). Significant advances were made in understanding molecular mechanisms linking FFA with insulin resistance: ranging from mechanistic substrate competition between FFA oxidation and glucose utilization with allosteric inhibition of glycolytic pathway enzymes to accumulation of several lipid-based intermediates with profound intracellular regulatory functions, such as LCFA-CoA (long-chain fatty acid-coenzyme A) and activation of specific isoforms of protein-kinase C (isoforms β, δ and θ) which subsequently phosphorylates several intracellular proteins including a key element in insulin receptor-mediated signal transduction, IRS-1 (insulin receptor substrate).

Lifestyle interventions (regular physical activity and dietary intervention) play a central role in the management of obesity, livers steatosis and Type 2 diabetes by multiple mechanisms, including reduction in spontaneous adipose tissue lipolysis. Human studies demonstrated decreased lower spontaneous lipolysis in active compared to sedentary subjects and decreased lipolytic rate was reported after 3-month exercise training and diet-induced weight loss. Molecular mechanisms mediating decreased lipolysis include improved sensitivity of adipocytes to insulin, a major anti-lipolytic hormone, as well as increased sensitivity to anti-lipolytic α2-adrenergic effect of circulating catecholamines. Importantly, using adipose tissue microdialysis technique, the investigators observed reduced α2-adrenergic signaling in diabetic subjects with severe OSA, opening a rationale for exercise-based interventions to reduce lipolysis in OSA. However, future research focusing on mechanisms behind dysregulated adipose tissue lipolysis in OSA is needed, as hypoxia (characteristic for OSA) directly induces multiple transcriptional and mitochondrial changes in adipocytes stimulating lipolysis in vitro and no studies evaluated whether adipose tissue lipolysis (including α2/β2 adrenergic signaling balance) can in fact be modified by lifestyle interventions in subjects with OSA. Besides beneficial metabolic effects of lifestyle-induced weight loss, adiposity reduction in the whole body and subsequent reduction in tongue / parapharyngeal tissue volume helps to keep airways opened during sleep (reducing the severity of OSA) and helps to better tolerate CPAP treatment (less external positive pressure required to keep airways opened). Lifestyle intervention thus induces additional beneficial effects, independent of molecular changes in adipose tissue and liver.

ELIGIBILITY:
Inclusion Criteria:

* mild (AHI < 10) or severe (AHI > 30) OSA diagnosed by home sleep study
* BMI 30-40 kg/m2
* age 18 - 65 years
* absence of diabetes mellitus (fasting glucose level < 7 mmol/l, HBA1c < 48 mmol/l and oGTT < 11.1 mmol/L 2 hours after 75g oral glucose load)
* no treatment with drugs affecting lipolysis (betablockers, alpha adrenergic blockers, glucocorticoids).

Exclusion Criteria:

* cardiac, renal or respiratory; chronic inflammatory or cancer disease
* body weight change more than 5 kg in last 3 months
* inability to participate in the life-style program
* inability to give an informed consent
* participation in another research project
* pregnancy or planned pregnancy during the study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Glycerol release (lipolysis) in adipose tissue measured by microdialysis | Baseline and 6 months
  Changes in interstitial glycerol concentration in adipose tissue before and after exercise and dietary intervention

SECONDARY OUTCOMES:
Weight loss measurements | 6 months
  5-10% weight loss by exercise and dietary intervention

CONTACTS AND LOCATIONS:
Overall Officials: Jan Polak, MD, PhD, Principal Investigator — Vascular surgery, University hospital Královské Vinohrady, Prague
Locations (1):
- University Hospital Královské Vinohrady, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No